CLINICAL TRIAL: NCT05000047
Title: 3D Ear Scanner-Workflow Timing and Preferences Compared to Traditional Silicone Earmold Impressions
Brief Title: Clinical Performance Evaluation of 3D Ear Canal Scanning Technology
Status: Completed | Type: Observational
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Other Study IDs: SRF-371
Record Dates: First submitted 2021-06-09; First posted 2021-08-11 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Ear Mold Impression Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- All participants: All study participants who have bilateral earmold impressions completed using both a 3D ear scanner and the conventional procedure using silicone impression material.
  Interventions: Device: 3D ear scanner; Other: Conventional silicon ear impressions

INTERVENTIONS:
Device: 3D ear scanner — A commercially-available ear scanning device used according to standard of care. A hand-held device is used and is considered less invasive than conventional earmold impressions.
Other: Conventional silicon ear impressions — A two part silicon impression material that is used to fill the ear and produce a physical cast of the ear canal. The procedure is standard of care.

SUMMARY:
Study participants will undergo ear canal impressions in a standard of care protocol utilizing two methodologies: 3D ear scanning using a commercially-available ear scanning device, and conventional silicone impression material. The elapsed time of each procedure will be captured for each participant, and the average duration of the two methodologies will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Hearing impairment (any degree, type, and configuration)

Exclusion Criteria:

* Absent or abnormal external auditory canal and/or external auditory meatus.
* Positive history of external/middle ear surgery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with anatomically typical external auditory canals/meatus who have any degree, type, and configuration of hearing impairment.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Seitz-Paquette, Principal Investigator — Sonova USCS
Locations (1):
- Phonak Audiology Research Center, Aurora, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 30 enrolled participants, 30 met inclusion criteria and completed the study.
Groups:
- All Participants: All participants who have bilateral impressions taken with both methodologies.
  1. A commercially-available ear scanning device used according to standard of care. A hand-held device is used and is considered less invasive than conventional earmold impressions.
  2. A two part silicon impression material that is used to fill the ear and produce a physical cast of the ear canal. The procedure is standard of care.
Period: Overall Study
Arm/Group | All Participants
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who have bilateral impressions taken with both methodologies.
  1. A commercially-available ear scanning device used according to standard of care. A hand-held device is used and is considered less invasive than conventional earmold impressions.
  2. Conventional silicon ear impressions: A two part silicon impression material that is used to fill the ear and produce a physical cast of the ear canal. The procedure is standard of care.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] — Age range from 40 to 88 years, with a mean age of 71.4 years.
  years | 71.4 [40 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Elapsed Time in Minutes to Complete Bilateral Ear Impressions
Description: The total time in minutes, required for sub-investigators to complete each impression methodology on each participant, according to a standard of care procedure . For the silicone impressions, time was started after otoscopy and cerumen management of both ears, and just before prepping and placing the otoblocks. The timer stopped after the audiologist was satisfied with both ear impressions and placed them in box. For the ear scan, time was started after otoscopy of both ears, and just before prepping the headset and hand-held scanner. The timer stopped after the 3D scan was reviewed for each ear and audiologist satisfied with result. The time reported is how long it took for clinician to finish one complete set of impressions, which included a right and a left ear impression. Separate times for each ear was not recorded.
Time Frame: Day one
Population: All earmold impression sets (right ear, left ear) that were taken by sub-investigator using both silicone and 3D scanning technologies.
Measure: Mean (Full Range); unit: Minutes
Units Other Than Participants: Set of earmold impressions
Groups:
- Set of Ear Impressions Taken Using 3D Scanner: Set (right ear, left ear) of impressions completed via a commercially available 3D ear scanner, which is used according to standard of care.
- Set of Impressions Taken Using Traditional Silicone Ear Impression Material and Technique: Set (right ear, left ear) of impressions taken using a two part silicon impression material which fills the ear and produces a physical cast of the ear canal. The procedure is standard of care.
Arm/Group | Set of Ear Impressions Taken Using 3D Scanner | Set of Impressions Taken Using Traditional Silicone Ear Impression Material and Technique
Number analyzed (Participants) | 30 | 30
Number analyzed (Set of earmold impressions) | 30 | 30
Minutes | 8.15 [5.55 to 14.4] | 6.28 [5.75 to 8.73]

2. Secondary Outcome: Subjective Feedback of Overall Experience of Both Ear Impression Procedures
Description: Each participant answered the question "How do you rate your experience of the recently performed ear canal impression/scanning?" after each procedure. Participants rated their overall experience on a scale from 1 (worst) to 5 (best).
Time Frame: Day one
Population: All participants who have both silicone and scanned ear impressions completed
Measure: Mean (Full Range); unit: score on a scale
Groups:
- 3D Scanning Technology: All participants who have bilateral impressions completed using a commercially available 3D ear scanner, used according to standard of care.
- Conventional Silicone Impression Procedure: All participants who have bilateral impressions completed using a two part silicon impression material which fills the ear and produces a physical cast of the ear canal. This procedure is done according to standard of care.
Arm/Group | 3D Scanning Technology | Conventional Silicone Impression Procedure
Number analyzed (Participants) | 30 | 30
score on a scale | 4.6 [2 to 5] | 3.9 [1 to 5]

3. Secondary Outcome: Subjective Feedback, Pleasantness of Experience
Description: Each participant answered the question "How pleasant do you rate the impression/scanning procedure?" after each procedure. Participants rated the the pleasantness on a scale from 1 (very pleasant) to 5 (very unpleasant).
Time Frame: Day one
Population: All participants who had both silicone and scanned ear impressions completed
Measure: Mean (Full Range); unit: score on a scale
Groups:
- 3D Scanning Technology: All participants who have bilateral impressions taken via a commercially available 3D ear scanner. This is done according to standard of care.
- Conventional Silicone Impression Procedure: All participants who have bilateral impressions taken using a two part silicone impression material which fills the ear and produces a physical cast of the ear canal. This is performed according to standard of care.
Arm/Group | 3D Scanning Technology | Conventional Silicone Impression Procedure
Number analyzed (Participants) | 30 | 30
score on a scale | 1.73 [1 to 3] | 2.4 [1 to 4]

4. Secondary Outcome: Subjective Feedback on the Perceived Improvement of Actual Device Fitting Using Each Impression Procedure Compared to a Non-custom Hearing Aid Fitting
Description: Each participant answered the question at the end of each procedure- "Compared to a non-custom fitting, do you feel that the method of impression/scanning improves the hearing aid process for you?", and rated on a scale from 1 (very improved) to 5 (much worse).
Time Frame: Day one
Population: All participants who had both silicone and scanned ear impressions completed
Measure: Mean (Full Range); unit: score on a scale
Groups:
- 3D Scanning Technology: All participants who have bilateral impressions completed using a commercially available 3D ear scanner. This is performed according to standard of care.
- Conventional Silicone Impression Procedure: All participants who have bilateral impressions taken using a two part silicone impression material which fills the ear and produces a physical cast of the ear canal. This is done according to standard of care.
Arm/Group | 3D Scanning Technology | Conventional Silicone Impression Procedure
Number analyzed (Participants) | 30 | 30
score on a scale | 1.77 [1 to 3] | 2.13 [1 to 4]

5. Secondary Outcome: Sub-investigator Clinician Subjective Rating of Ease of Procedure on a Scale From 1 (Not at All Easy) to 10 (Most Ease)
Description: Sub-investigators answered a question after each procedure on each participant- "How easy was it to perform the procedure? on a scale from 1 (not at all easy) to 10(most ease).
Time Frame: Day 1
Population: All earmold impression sets (right ear, left ear) that were taken by sub-investigators using both silicone and 3D scanning technologies. Sub-investigators were not considered enrolled but contributed to this assessment.
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: set of earmold impressions
Groups:
- 3D Scanning Technology: Set (right ear, left ear) of impressions completed via a commercially available 3D ear scanner. The procedure is standard of care.
- Conventional Silicone Impression Procedure: Set (right ear, left ear) of impressions taken using a two part silicon impression material which fills the ear and produces a physical cast of the ear canal. The procedure is standard of care.
Arm/Group | 3D Scanning Technology | Conventional Silicone Impression Procedure
Number analyzed (Participants) | 30 | 30
Number analyzed (set of earmold impressions) | 30 | 30
score on a scale | 8.13 [2 to 10] | 9.27 [4 to 10]

6. Secondary Outcome: Sub-investigator Clinician Subjective Rating of Individual Potential for Improvement When Performing Each Procedure 1 (no Potential for Improvement) to 3 (a Lot of Potential for Improvement)
Description: Sub-investigators answered a question after each procedure on each participant they saw- "Do you feel like there was any potential for improvement when performing this procedure?". Each sub-investigator rated their own potential for improvement on a scale from 1(no potential for improvement, clinician was very satisfied with impression) to 3 (a lot of potential for improvement, clinician felt impression was inferior).
Time Frame: Day 1
Population: All earmold impression sets (right ear, left ear) that were taken by clinician using both silicone and 3D scanning technologies. Sub-investigator clinicians were not considered enrolled but did contribute to this assessment.
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: set of earmold impressions
Groups:
- 3D Scanning Technology: Set (right ear, left ear) of impressions completed via a commercially available 3D ear scanner, which is used according to standard of care.
Arm/Group | 3D Scanning Technology | Conventional Silicone Impression Procedure
Number analyzed (Participants) | 30 | 30
Number analyzed (set of earmold impressions) | 30 | 30
score on a scale | 1.6 [1 to 3] | 1.2 [1 to 2]

7. Secondary Outcome: Sub-investigator Clinician Subjective Rating of Individual Confidence That Method of Impression Will Yield a Quality Custom Product for the Participant on a Scale From 1 (Not at All Confident) to 3 (Very Confident).
Description: Sub-investigators answered a question after each procedure on each participant they saw- "How confident are you that the method of impression/scanning will yield a quality custom product?" on a scale from 1 (not at all confident) to 3 (very confident).
Time Frame: Day 1
Population: All earmold impression sets (right ear, left ear) that were taken by clinician using both silicone and 3D scanning technologies. Clinicians were not considered enrolled but did contribute to this assessment.
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: set of earmold impressions
Groups:
- 3D Scanning Technology: Set (right ear, left ear) of impressions taken using the 3D scanner. The procedures is standard of care.
Arm/Group | 3D Scanning Technology | Conventional Silicone Impression Procedure
Number analyzed (Participants) | 30 | 30
Number analyzed (set of earmold impressions) | 30 | 30
score on a scale | 2.6 [1 to 3] | 2.9 [2 to 3]

8. Secondary Outcome: Clinician Subjective Rating of Overall Experience of Each Procedure.
Description: Clinicians answered a question after each procedure on each participant they saw- "How would you rate the overall experience of performing this procedure?" using a scale from 1 (worst) to 5 (best).
Time Frame: Day 1
Population: as for outcome 7
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: Earmold impression sets
Groups:
- 3D Scanning Technology: Set (right ear, left ear) of impressions taken using the 3D scanner. The procedure is standard of care.
- Conventional Silicone Impression Procedure: Set (right ear, left ear) of impressions taken using conventional silicone material. The procedure is standard of care.
Arm/Group | 3D Scanning Technology | Conventional Silicone Impression Procedure
Number analyzed (Participants) | 30 | 30
Number analyzed (Earmold impression sets) | 30 | 30
score on a scale | 4.2 [2 to 5] | 4.5 [3 to 5]

ADVERSE EVENTS:
Time Frame: up to 30 days after participant was seen for impressions.
Description: Any adverse events that occur at time of appointment are documented on adverse event template form (TPL-518) and follow up continues with participant for 30 days or until event is resolved, or a referral has been made to appropriate medical professional.
Groups:
- All Participants: All participants will have bilateral impressions taken with both methodologies.
  1. A commercially-available ear scanning device used according to standard of care. A hand-held device is used and is considered less invasive than conventional earmold impressions.
  2. Conventional silicon ear impressions: A two part silicon impression material that is used to fill the ear and produce a physical cast of the ear canal. The procedure is standard of care.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT05000047/Prot_SAP_000.pdf